CLINICAL TRIAL: NCT06448871
Title: Usefulness of Ultrasound to Assess Sarcopenia in Individuals With Prader Willi Syndrome
Brief Title: Ultrasound to Assess Sarcopenia in Prader Willi Syndrome
Acronym: PWS
Status: Completed | Type: Observational
Sponsor: Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: TCRD-TPE-112-28
Record Dates: First submitted 2024-05-02; First posted 2024-06-07 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-09

CONDITIONS: Prader-Willi Syndrome; Sarcopenia; Metabolic Syndrome
Keywords: Prader-Willi Syndrome; Sarcopenia; Ultrasound; skeletal muscle; body composition
MeSH Terms: conditions — Prader-Willi Syndrome; Sarcopenia; Metabolic Syndrome | interventions — Absorptiometry, Photon

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — No biospecimen will be used in this study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- group 1, pws group: Individuals with PWS, aged 7 to 65 years, and able to follow simple instructions in chinese language.
  Interventions: Diagnostic Test: Ultrasound assessment of the right lower extremity muscles; Diagnostic Test: Dual-energy X-ray absorptiometry (DXA) scan

INTERVENTIONS:
Diagnostic Test: Ultrasound assessment of the right lower extremity muscles — Rectus femoris cross sectional area (RFCSA), RF muscle thickness, vastus lateralis (VL) muscle thickness, Gastrocnemius medialis (GM) muscle thickness, VL pennation angle (PA), and GM PA.
Diagnostic Test: Dual-energy X-ray absorptiometry (DXA) scan — skeletal muscle mass (SM), appendicular skeletal muscle mass index (ASMI), total lean body mass (LBM), total fat mass (BF), percentage fat mass, and fat mass index (FMI).

SUMMARY:
The aim of the study is to examine the clinical applicability of ultrasound as a diagnostic tool for sarcopenia in individuals with PWS by investigating the association between ultrasound-derived measurements, DXA-derived measurements, and sarcopenia-related outcomes.

DETAILED DESCRIPTION:
Sarcopenia is an age-related loss of muscle mass plus low muscle strength, and/or low physical performance, that may affect over 25% of individuals over the age of 60, resulting in an increased likelihood of developing disability. Abnormal body composition with an increased in body fat mass and a decreased in skeletal muscle mass were noted in individuals with Prader Willi syndrome (PWS), thought to be related to hormonal deficiencies due to hypothalamic dysfunction, presenting as a unique congenital model of sarcopenia.

Muscle mass can be measured by dual-energy X-ray absorptiometry (DXA) scan device, but it is expensive, increased radiation exposure, and not easily accessible in all clinical practice. Ultrasound (USD) is a non-invasive, without ionising radiation, low-cost, and easily accessible tool for the assessment of soft tissue. There were increasing evidence for the use of USD in the measurement of muscle thickness (MT), cross-sectional area (CSA) and pennate anle (PA) of different muscle groups in different populations. However, the use of USD as a routine diagnostic tool in individuals with PWS has not been reported yet.

The aim of the study is to examine the clinical applicability of ultrasound as a diagnostic tool for sarcopenia in individuals with PWS by investigating the association between ultrasound-derived measurements, DXA-derived measurements, and sarcopenia-related outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Genetically diagnosed individuals with PWS who can cooperate with the examinations

Exclusion Criteria:

* Individuals with PWS who have arthritis, fractures, or severe musculoskeletal deformities that could interfere with the examinations.
* Individuals with PWS who have severe cognitive impairment and are unable to read or sign the written consent.

Ages: 7 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All individuals with genetically confirmed PWS will be recruited from one of the Northern hospital outpatient center in Taiwan in the given time period.
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2022-10-17 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Muscle thickness ultrasound | 1 day
  Ultrasound scanning of the muscle thickness of rectus femoris (RF), vastus lateralis (VL), and gastrocnemius medialis (GM) using B-mode ultrasonography (LOGIQ S8, GE Healthcare, USA) and a 7-15 MHz linear array transducer.
Cross-sectional area ultrasound | 1 day
  Ultrasound scanning of the cross sectional area of rectus femoris (RF) using B-mode ultrasonography (LOGIQ S8, GE Healthcare, USA) and a 7-15 MHz linear array transducer.
Pennation angle ultrasound | 1 day
  Ultrasound scanning of the pennation angles of vastus lateralis (VL) and gastrocnemius medialis (GM) using B-mode ultrasonography (LOGIQ S8, GE Healthcare, USA) and a 7-15 MHz linear array transducer.
DXA: total lean body mass | 1 day
  Lean index of total lean body mass (LBM) with Hologic QDR-4500A, Hologic, Inc., Waltham, MA, USA
DXA: skeletal muscle (SM) | 1 day
  Lean index of skeletal muscle (SM) with Hologic QDR-4500A, Hologic, Inc., Waltham, MA, USA
DXA: appendicular skeletal muscle mass index (ASMI) | 1 day
  Lean index of appendicular skeletal muscle mass index (ASMI) with Hologic QDR-4500A, Hologic, Inc., Waltham, MA, USA
DXA: fat mass index (FMI) | 1 day
  Adipose index of fat mass index using Hologic QDR-4500A, Hologic, Inc., Waltham, MA, USA.
DXA: body fat mass (BFM) | 1 day
  Adipose index of body fat mass (BFM) using Hologic QDR-4500A, Hologic, Inc., Waltham, MA, USA.
DXA: percentage fat mass | 1 day
  Adipose index of percentage fat mass using Hologic QDR-4500A, Hologic, Inc., Waltham, MA, USA.

SECONDARY OUTCOMES:
Handgrip and lateral pinch strength | 1 day
  Grip strength and lateral pinch will be assessed bilaterally using an isometric Baseline hydraulic hand dynamometer and pinch gauge.
Physical performance test: SPPB | 1 day
  The short physical performance battery (SPPB) will be used, which measures balance, walking speed, strength, and endurance in the lower limbs, and is scored from zero to 12 (worst to best score).
Physical performance test: gait speed | 1 day
  In the gait speed test participants walk over a 4-meter distance at their normal pace.
Physical performance test: five-time chair stand test | 1 day
  In the 5-time chair stand test participants perform five sit-to-stand movements as quickly as possible

CONTACTS AND LOCATIONS:
Overall Officials: Valeria Chiu, MD, Principal Investigator — Taichung Tzu Chi Hospital
Locations (1):
- Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No